CLINICAL TRIAL: NCT06933446
Title: Effect of Release of Trigger Points on Functional Capacity, Biomechanical and Physiological Variables in Recovery After Game Simulation in Water Polo Athletes
Brief Title: Effect of Myofascial Release on Post-Exercise Recovery in Water Polo Athletes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luis Gustavo Lizi Jorge (Other)
Responsible Party: Sponsor-Investigator, Luis Gustavo Lizi Jorge, Physiotherapist, Universidade do Sagrado Coração
Organization: Universidade do Sagrado Coração (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 6.711.962
Record Dates: First submitted 2025-03-26; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Fatigue
Keywords: fatigue; physical exertion; post-exercise recovery
MeSH Terms: conditions — Fatigue | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myofascial Release (Active Comparator)
  Interventions: Other: Classic Massage
- Classic Massage (Placebo Comparator)
  Interventions: Other: Myofascial Release

INTERVENTIONS:
Other: Myofascial Release — A myofascial release protocol, applied to the thigh muscles in post-effort recovery in water polo athletes.
  Arms: Classic Massage
Other: Classic Massage — Massagem clássica, com pressão superficial, utilizada para atingir apenas tecidos subcutâneos, sem que haja ação sobre músculos e fáscias
  Arms: Myofascial Release

SUMMARY:
Objective: To assess the acute effect of a myofascial release protocol applied to the adductor muscles of the thigh on functional, biomechanical, and physiological variables. Methods: This study is a randomized, double-blind, two-arm crossover clinical trial that will analyze male water polo athletes aged 16 to 25 years recruited from a sports training center in the city of Bauru. Data related to the following parameters will be collected for the physical evaluation: functional performance, through the jump test; biomechanical, through maximum isometric torque of hip adductors, electromyography of the hip and gluteus medius muscles; and physiological, through the analysis of serum markers of muscle damage and inflammation, and heart rate variability. After the initial evaluation, the participants will be randomly divided into two groups: intervention group and sham group. Then, all participants will perform a game simulation. After the game, the participants will receive the intervention designated for each group. For the intervention group, a manual therapy protocol will be applied, based on myofascial release in the thigh region that presents trigger points. For the Sham group, a manual technique, called classic massage, will be applied, with superficial pressure, used to reach only subcutaneous tissues, without acting on muscles and fascia. This protocol will be repeated at four different times, always after the games. After a washout week, the participants will change groups and the data collection protocol will be applied again.

ELIGIBILITY:
Inclusion Criteria:

1. Male athletes;
2. Age 16 to 25 years old;
3. Have at least one year of experience in the sport;
4. Perform a training load of at least 10 hours per week in the sport;
5. Participate in at least regional level competitions

Exclusion Criteria:

1. Have no reports of muscle injury in the thigh in the three months prior to the study,
2. Joint injuries in the hip, such as femoroacetabular impingement or tendinopathies of the tendons of the hip muscles or trochanteric, iliopectineal or ischial bursitis diagnosed by a clinician;
3. Do not present a drop in -performance for more than four weeks that could characterize the occurrence of non-functional overreaching or signs of overtraining syndrome

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male athletes, age 16 to 25 years old, have at least one year of experience in the sport
Enrollment: 16 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Vertical Jump Test | From enrollment to the end of treatment at 2 weeks
Maximum Voluntary Isometric Torque of the Hip Adductors | From enrollment to the end of treatment at 2 weeks
Electromyography of Adductors, Gluteus Medius and Transversus Abdominis | From enrollment to the end of treatment at 2 weeks
Collection of Serum Markers | From enrollment to the end of treatment at 2 weeks
  The markers: creatine kinase (CK; Units of Measure= U/L), lactate dehydrogenase (LDH; Units of Measure= UI/L), myoglobin (Myo; Units of Measure= ng/mL), erythrocyte sedimentation rate (ESR; Units of Measure= mm/h), tumor necrosis factor alpha (TNFA; Units of Measure= Å) will be considered for analysis of muscle damage markers and will be determined through specific kits and following the manufacturer's instructions.
Heart Rate Variability | From enrollment to the end of treatment at 2 weeks
  Heart rate variability (HRV) will be collected, at rest, through a non-invasive method used to measure cardiac autonomic control, to assess the autonomic nervous system (ANS), and the RR interval will be recorded by a portable heart rate monitor.

SECONDARY OUTCOMES:
Effort Control Variables: Subjective Perception of Exertion and Lactate Threshold | From enrollment to the end of treatment at 2 weeks
  To estimate the intensity of the exercise, the method proposed by Foster (1998) will be used, which suggests multiplying the subjective perception of exertion (RPE) of the session by the total duration of the training session (sRPE), with the results expressed in arbitrary units (u.a.). To quantify performance during the game, lactate will be collected at the end of each quarter of the game, through blood collections from the earlobe (25 μL) to analyze the peak lactate concentration ([La-]peak) of the effort.

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca Gasparoto Carmezin, Acadêmica em Fisioterapia, Principal Investigator — Universidade do Sagrado Coração
Locations (1):
- Universidade do Sagrado Coração, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No